CLINICAL TRIAL: NCT07214948
Title: An Open, Parallel-group, Randomized, Early Feasibility Trial to Evaluate the Initial Safety and Performance of the INGA Catheter in Labor Induction
Brief Title: Open, Randomized Feasibility Trial on the Safety and Performance of the INGA Catheter for Labor Induction
Acronym: INGA-RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalto University (Other)
Collaborators: University of Mississippi Medical Center (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00089090; ARPA-H-ICHUB-24-101-1675/SWH-2 (Other Grant/Funding Number: ARPA-H)
Record Dates: First submitted 2025-10-01; First posted 2025-10-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Induction of Birth; Cervical Ripening; Cervical Ripening and Induction of Labor
Keywords: Induction of labor; Balloon Catheter; Cervical ripening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- INGA Catheter (Experimental)
  Interventions: Device: INGA Catheter
- Currently used induction catheter (Other): Insertion of the currently used induction balloon catheter through the cervical canal into the uterus is performed for labor induction. During a vaginal examination, the Investigator inserts the catheter so that the balloon tip lies between the amniotic membranes and the internal cervical os. The balloon is filled with 50-75 ml of sterile saline (NaCl) and secured to the upper thigh to maintain gentle traction. The catheter remains in place for up to 24 hours or until spontaneous expulsion. If not expelled, it is removed after 24 hours.
  After expulsion or removal, cervical status and Bishop score are assessed. If Bishop ≥ 6, amniotomy and/or oxytocin induction are initiated within one hour. If Bishop < 6, further management follows
  Interventions: Device: Currently used single balloon catheter

INTERVENTIONS:
Device: INGA Catheter — Insertion of the INGA balloon catheter (medical device) through the cervical canal into the uterus is performed for labor induction. During a vaginal examination, the Investigator inserts the catheter so that the balloon tip lies between the amniotic membranes and the internal cervical os. The balloon is filled with 50-75 ml of sterile saline (NaCl) and secured to the upper thigh to maintain gentle traction. The catheter remains in place for up to 24 hours or until spontaneous expulsion. If not expelled, it is removed after 24 hours.
  After expulsion or removal, cervical status and Bishop score are assessed. If Bishop ≥ 6, amniotomy and/or oxytocin induction are initiated within one hour. If Bishop < 6, further management follows
  Arms: INGA Catheter
Device: Currently used single balloon catheter — Insertion of a balloon catheter through the cervical canal into the uterus for induction of labor.
  Arms: Currently used induction catheter

SUMMARY:
This study investigates the safety and usability of the new INGA catheter for labor induction.

Labor induction is common, with about one in three births being induced. In this study, the INGA catheter will be compared to a currently used method. The INGA catheter is a single-balloon device that works similarly to a Foley catheter but is made from different materials. Feedback will be collected from both healthcare professionals and participating women.

DETAILED DESCRIPTION:
Screening Phase

Before any study-related procedures are initiated, participants will be asked to read and sign the informed consent form. Once consent is obtained, the following screening assessments will be performed to determine eligibility for participation:

* Confirmation of informed consent.
* Review of inclusion and exclusion criteria to ensure suitability for the study.
* Collection of medical and demographic information, including medical history, concurrent or previous medications, planned delivery date, gestational age, and indication for labor induction.
* Cervical assessment by palpation.
* Measurement of blood pressure and heart rate.
* Cardiotocography (CTG) monitoring of fetal heart rate and uterine contractions for a minimum of 30 minutes.
* Ultrasound examination within one week prior to induction, to evaluate fetal weight, well-being, and overall status.

If the screening assessments confirm that the participant meets all eligibility criteria, she will proceed to the study phase and receive the assigned study device.

Study Device and Randomization

After signing the informed consent form, each eligible participant will be randomly assigned to one of two treatment groups:

* 1 in 3 chance of receiving the commonly used balloon catheter for labor induction.
* 2 in 3 chance of receiving the INGA catheter, the investigational device being studied.

This is an open-label study, meaning that both the participant and the study personnel (including the investigator and sponsor) will know which device is used.

The study procedure follows the standard clinical process for balloon catheter-based induction of labor. No additional or experimental procedures are performed beyond the use of the assigned catheter. The only difference from routine clinical practice is the use of the INGA catheter in the investigational group.

Study Procedures

Participants will undergo the following procedures as part of the study:

* The catheter (either the standard or INGA catheter) will be inserted by a trained physician through the vagina and advanced through the cervical canal.
* The balloon portion of the catheter will be inflated with sterile saline to secure its position and will be fastened to the inner thigh to maintain placement.
* Fetal heart rate monitoring (CTG) will be performed both before and after catheter placement, following standard hospital protocol.
* Cervical ripeness will be assessed prior to catheter insertion and again after catheter removal or spontaneous expulsion.
* The catheter will remain in place until it detaches spontaneously or for a maximum duration of 24 hours.
* After catheter removal, cervical status will be reassessed, and labor induction will continue according to the hospital's standard of care.

Throughout the procedure, the principal investigator and hospital staff will closely monitor the induction process and ensure the safety and well-being of both the mother and the fetus.

Comprehensive data will be collected on:

* The course of pregnancy and labor induction process.
* Delivery outcomes, including type and duration of delivery.
* Maternal safety data, including any adverse events or complications. Infant Assessments

Following labor and delivery, the following evaluations will be conducted for the newborn:

* Birth weight and length.
* Apgar score at 5 minutes post-delivery.
* Collection of clinical data related to any neonatal diagnoses, treatments, or medical conditions.

Questionnaires

To assess user experience and device tolerability, the following questionnaires will be completed:

* Participants will be asked to complete a short questionnaire evaluating their overall comfort, well-being, and any discomfort or pain experienced during placement and use of the balloon catheter.
* The physician performing the catheter placement will complete a usability questionnaire to assess the practicality, ease of use, and general handling of the device.

Post-Treatment Phase

After completion of the study procedure:

* The study device (INGA catheter or standard catheter) will be used only during this research study and will not be available for use after study participation ends.
* No additional study visits or treatments are required once labor induction and delivery are complete.
* Routine post-delivery care will be provided according to standard hospital practices.

Participant Expectations

By agreeing to participate in this study, each participant is expected to:

* Read, understand, and sign the informed consent document.
* Meet all inclusion criteria and not meet any exclusion criteria.
* Understand that randomization will determine which study device is used.
* Allow collection of maternal and neonatal health data for study analysis.
* Complete the participant questionnaire regarding her experience with the catheter.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged ≥18 and ≤56 years
* An unripe cervix, ≤6 points according to the Bishop score assessment (0-10-point scale)
* Planned induction of labor by balloon catheter method
* Gestational age at the time of the study ≥ 37 weeks (gestational age confirmed by ultrasound before the 21st week of pregnancy)
* Singleton pregnancy
* Cephalic presentation
* The subject understands the study information and signs the informed consent

Exclusion Criteria:

* Preterm induction of labor (<37 weeks of gestation)
* Abnormal Cardiotocography (CTG) at inclusion
* Spontaneous rupture of membranes at inclusion
* Clinically significant vaginal bleeding with a need of hospitalization in the third trimester
* Clinical active vaginal or uterine infection
* Maternal Human Immunodeficiency Virus (HIV), hepatitis C, or hepatitis B
* Uterine scar (including previous cesarean section)
* Condition requiring immediate delivery of the fetus or mother
* Presence of eclampsia
* Severe Preeclampsia [Blood pressure (BP)≥ 160/110 and any of the following: thrombocytopenia with platelet count <100 × 10e9/L, HELLP- syndrome ( Hemolysis, Elevated Liver enzymes and Low Platelets), progressive renal insufficiency, pulmonary edema ]
* Severe fetal growth restriction (Fetal Growth Restriction (FGR) fetal growth <-2 SD/<10th percentile)
* Estimated fetal weight ≥ 2 Standard Deviation /≥ 95th percentile
* Reduced amniotic fluid volume (deepest vertical pocket <30 mill meter)
* Breech or transverse fetal position
* Multiple pregnancy
* Vasa previa or placenta previa
* Umbilical cord prolapses
* Bishop score ≥6 on cervical assessment prior to labor induction
* Receiving epidural anesthesia prior to catheter insertion
* Refusal to participate in the study and/or insufficient language skills to understand the study information and/or consent form

Ages: 18 Years to 56 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 90 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Bishop Score Change | From catheter insertion to detachment
  Change in Bishop score (A scale from 1 to 10) during cervical ripening, with scores assessed before catheter insertion and after catheter detachment.

SECONDARY OUTCOMES:
Placement success | At catheter insertion
  Whether the catheter is placed successfully
Retention time of balloon catheter | From catheter placement to detachment, 0-24 hours
  The time the balloon catheter remains in the cervix for cervical ripening
Induction to delivery interval | rom the start of balloon catheter insertion until the birth of the neonate, 0-48 hours
  Time from initiation of labor induction (balloon catheter insertion) to the delivery of the neonate. This includes both the cervical ripening phase and active labor. The outcome will capture the total duration of the induction-to-delivery process.
Mode of delivery | From enrolment to birth
  The type of delivery for the participant, categorized as vaginal, vaginal operative or cesarean delivery
Pain experience during catheter insertion and in-place time | Within 60 minutes from catheter insertion
  The participants will complete a structured questionnaire to assess any potential pain experienced during catheter placement and retention
Professional's experience of catheter insertion and usability | From catheter insertion to detachment
  The Investigators will complete a structured questionnaire to evaluate the ease of catheter placement, usability, quality, appearance, and balloon inflation. The questionnaire also includes questions regarding their willingness to use technological applications in the context of labor induction.

CONTACTS AND LOCATIONS:
Overall Officials: Leena Rahkonen, MD,PhD, Associate Professor, Study Chair — Aalto University

IPD SHARING:
Plan to Share IPD: Undecided